CLINICAL TRIAL: NCT07266467
Title: Efficacy and Safety of Leymovir Versus Valganciclovir in Prevention of Cytomegalovirus Infection and Cytomegalovirus Disease in Chinese Kidney Transplant Recipients
Acronym: CAPS01
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Chinese People's Liberation Army Northern Theater Command General Hospital (Unknown); The First Hospital of Jilin University (Other); The Affiliated Hospital of Qingdao University (Other); Qianfo Mountain Hospital, Shandong Province (Unknown); The First Affiliated Hospital of Anhui Medical University (Other); Eastern Theater General Hospital (Unknown); Shu lan Hospital (Unknown); Shanghai Zhongshan Hospital (Other); Tongji Hospital (Other); The Second Xiangya Hospital, Central South University (Unknown); The First Affiliated Hospital of Zhengzhou University (Other); Second Affiliated Hospital of Guangzhou Medical University (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Beijing Chao Yang Hospital (Other); RenJi Hospital (Other); Nanfang Hospital, Southern Medical University (Other); Tsinghua Changgeng Hospital, Beijing (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: XJTUAF2025-CAPS01
Record Dates: First submitted 2025-05-11; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-03

CONDITIONS: Kidney Transplant
Keywords: Kidney Transplant; cytomegalovirus; letemovir; valganciclovir; Randomized control
MeSH Terms: interventions — letermovir; Valganciclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Valganciclovir (Experimental): Experimental drug: Valganciclovir. Dose: 450mg. Dosing interval: once daily. Route of administration: oral. Course of treatment: Starting within 7 days (random day) after kidney transplantation and continuing until the 14th week (about 100 days) after transplantation.
  Interventions: Drug: Valganciclovir
- Letermovir (Active Comparator): Drug name: Letermovir. Dose: 480mg. Dosing interval: once daily. Route of administration: oral. Course of treatment: Starting within 7 days (random day) after kidney transplantation and continuing until the 14th week (about 100 days) after transplantation.
  Interventions: Drug: Letermovir

INTERVENTIONS:
Drug: Letermovir — Drug name: Letermovir.
  Arms: Letermovir
Drug: Valganciclovir — Valganciclovir.
  Arms: Valganciclovir

SUMMARY:
the existing anti-CMV drugs mainly include valganciclovir, ganciclovir and foscarnet sodium, all of which act on DNA polymerase (pUL54), making them prone to cross resistance. DNA synthesis in normal cell is also catalyzed by DNA polymerase, which can also inhibit normal cell production, especially in metabolically active bone marrow cells, leading to bone marrow suppression. In addition, these drugs are mainly metabolized by the kidneys, causing damage to proximal renal tubular cells. Therefore, it is necessary to closely monitor the patient's renal function and adjust the dosage. Overall, the medical demand for effective and well-tolerated treatment methods for CMV infection management in kidney transplant recipients remains unmet, and safer anti-CMV drugs are urgently needed.

The target of letemovir is the CMV DNA terminal enzyme complex, which is different from the target of existing anti-CMV drugs, and does not exhibit cross resistance. Moreover, this target does not have a corresponding substance in mammalian cells and does not exhibit toxicity similar to DNA polymerase targets. In addition, letemovir is mainly metabolized by the liver, and urinary excretion can be ignored (<2% dose), so there is no need to adjust the dose according to renal function. Phase III registered clinical studies abroad have shown that letemovir is not inferior to valganciclovir in preventing CMV disease in kidney transplant recipients. Additionally, letemovir is safer and has a lower incidence of adverse reactions, especially leukopenia or granulocytopenia. However, there is still a lack of data on the use of kidney transplantation in Chinese population.

The aim of this study was to evaluate the efficacy and safety of letamovir in preventing CMV infection and CMV disease in kidney transplant recipients in China.

DETAILED DESCRIPTION:
the existing anti-CMV drugs mainly include valganciclovir, ganciclovir and foscarnet sodium, all of which act on DNA polymerase (pUL54), making them prone to cross resistance. DNA synthesis in normal cell is also catalyzed by DNA polymerase, which can also inhibit normal cell production, especially in metabolically active bone marrow cells, leading to bone marrow suppression. In addition, these drugs are mainly metabolized by the kidneys, causing damage to proximal renal tubular cells. Therefore, it is necessary to closely monitor the patient's renal function and adjust the dosage. Overall, the medical demand for effective and well-tolerated treatment methods for CMV infection management in kidney transplant recipients remains unmet, and safer anti-CMV drugs are urgently needed.

The target of letemovir is the CMV DNA terminal enzyme complex, which is different from the target of existing anti-CMV drugs, and does not exhibit cross resistance. Moreover, this target does not have a corresponding substance in mammalian cells and does not exhibit toxicity similar to DNA polymerase targets. In addition, letemovir is mainly metabolized by the liver, and urinary excretion can be ignored (<2% dose), so there is no need to adjust the dose according to renal function. Phase III registered clinical studies abroad have shown that letemovir is not inferior to valganciclovir in preventing CMV disease in kidney transplant recipients. Additionally, letemovir is safer and has a lower incidence of adverse reactions, especially leukopenia or granulocytopenia. However, there is still a lack of data on the use of kidney transplantation in Chinese population.

The aim of this study was to evaluate the efficacy and safety of letamovir in preventing CMV infection and CMV disease in kidney transplant recipients in China.

ELIGIBILITY:
Inclusion Criteria:

- 1) Age ≥18 years old, gender unlimited. 2) Receiving the first kidney transplant. 3) Be within 0 (ie, day of transplantation) to 7 days (inclusive) post-kidney transplant at the time of randomization.

4) Obtain informed consent signed .

Exclusion Criteria:

* 1)Received a previous solid organ transplant or HSCT. 2)Is a multi-organ transplant recipient (eg, kidney-pancreas). Note: Double kidney transplant recipients (ie, transplant of two kidneys from the same donor to the same recipient simultaneously) will be excluded.

  3)Has a history of CMV disease or suspected CMV disease within 6 months prior to randomization.

  4)Has evidence of CMV viremia at any time from the signing of the ICF or the transplant procedure until the randomization period; 5)Has suspected or known hypersensitivity to active or inactive ingredients of LET formulations, VGCV, GCV, formulations.

  6)Is on dialysis or plasmapheresis at the time of randomization. Note: For the purposes of this protocol, dialysis includes hemofiltration. Participant who: (1) has had dialysis or plasmapheresis within 7 days (inclusive) post-transplant but is not on dialysis or plasmapheresis at the time of randomization; and (2) is expected to remain off dialysis or plasmapheresis may be enrolled, provided that all other inclusion/exclusion criteria are met.

  7)Has post-transplant renal function of CrCI 10 mL/min at randomization (measured) locally). For this exclusion criterion, CrCl will be calculated using the Cockcroft-Gault equation using the most recently obtained and available serum creatinine value collected within 3 calendar days prior to and including the day of randomization and after the conclusion of any clinically warranted (at the discretion of the investigator) post-transplant dialysis or plasmapheresis.

  8)Has Child-Pugh Class C severe hepatic insufficiency at screening. 9)Has both moderate hepatic insufficiency AND moderate-to-severe renal insufficiency at screening.

Note: Moderate hepatic insufficiency is defined as Child-Pugh Class B. moderate-to-severe renal insufficiency is defined as CrCl <50 mL/min, as calculated by the Cockcroft-Gault equation, respectively.

10)Has any uncontrolled infection on the day of randomization. 11)Has documented positive results for human immunodeficiency virus antibody (HIV-Ab) test at any time prior to randomization, or for hepatitis C virus antibody (HCV-Ab) and with detectable HCV ribonucleic acid (RNA) within 90 days prior to randomization or hepatitis B surface antigen (HBsAg) within 90 days prior to randomization.

12)Requires mechanical ventilation, or is hemodynamically unstable, at the time of randomization.

13)Has a history of malignancy 5 years prior to signing informed consent except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer or carcinoma in situ; or is under evaluation for other active or suspected malignancy.

14)Is pregnant or expecting to conceive, is breastfeeding, or plans to breastfeed from the time of consent through at least 90 days following cessation of study therapy.

15)Has a history or current evidence of any condition, therapy, lab abnormality, or other circumstance that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or put the participant at undue risk, as judged by the investigator, such that it is not in the best interest of the participant to participate in this study.

16)laboratory value at screening: hemoglobin <8g/dL; Or neutrophils <1.0*109/L; Or platelet <25*109/L; Serum AST or ALT>5×ULN; Or serum total bilirubin >2.5×ULN; 17)Has received within 30 days prior to randomization or plans to receive during the study any of the following anti-CMV IgG antibody treatment or anti-CMV drug therapy including: Cidofovirb. CMV hyper-immune globulinc. Any investigational CMV antiviral agent/biologic therapy.

18)Has received within 7 days prior to randomization or plans to receive during the study any of the following anti-CMV drug therapy including: LET, GCV, VGCV, Foscarneth, ACV (at doses >3200 mg PO per day or >25 mg/kg IV per day), Valacyclovir (at doses >3 g PO per day), Famciclovir (at doses >1500 mg PO per day).

19)are expected to receive TCM or herbal treatment during study treatment and within 14 days after study administration; 20)Is currently participating or has participated in a study with an unapproved investigational compound or device within 28 days, or 5 x half-life of the investigational compound (excluding monoclonal antibodies), whichever is longer, of initial dosing on this study. Participants previously treated with an investigational monoclonal antibody will be eligible to participate after a 150-day washout period.

21)Has previously participated or is currently participating in any study involving administration of a CMV vaccine or another CMV investigational agent, or is planning to participate in a study of a CMV vaccine or another CMV investigational agent during the course of this study.

22)Is or has an immediate family member (eg, spouse, parent/legal guardian, sibling or child) who is investigational site or sponsor staff directly involved with this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of CMV disease at 52 weeks after transplantation | 52 weeks after transplantation
  Proportion of subjects diagnosed with CMV disease at week 52 after transplantation.

SECONDARY OUTCOMES:
Incidence of CMV disease at 14/24 weeks after transplantation | 14/24 weeks after transplantion
  Proportion of subjects diagnosed with CMV disease at week 14/26 after transplantation.
Time of CMV onset 52 weeks after transplantation | 52 weeks after transplantation
  From the day of transplant to the first diagnosis of CMV disease.
Incidence of CMV DNaemia at 14/26/52 weeks after transplantation | 14/24/52 weeks after transplantion
  Proportion of subjects diagnosed with CMV DNaemia at week 14/26/52 after transplantation.
Incidence and severity of all adverse events | 52 weeks after transplantation
  Proportion of subjects with any AE that occurred from the time the study intervention was assigned to 14 days after the study intervention was terminated. Saes will only be reported 14 days after stopping the study intervention until week 52 after transplantation.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Xi 'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No
Publish the statistical results after the completion of the experiment in the form of academic papers